CLINICAL TRIAL: NCT03911700
Title: Prospective, Multi-Center, Open-Label, Randomized, Controlled Trial of Phasix™ Mesh to Prevent Incisional Hernia Subsequent to Open Midline Laparotomy
Brief Title: Prophylactic Reinforcement of Ventral Abdominal Incisions Trial
Acronym: PREVENT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DVL-HE-018
Record Dates: First submitted 2019-04-04; First posted 2019-04-11 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Open Midline Laparotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Phasix™ Mesh (Experimental): Prophylactic onlay placement of mesh.
  Interventions: Device: Phasix™ Mesh
- Primary Suture Closure (No Intervention): Standard Fascial closure.

INTERVENTIONS:
Device: Phasix™ Mesh — Phasix™ Mesh is a resorbable mesh prepared from Poly-4-hydroxybutyrate (P4HB).
  Arms: Phasix™ Mesh

SUMMARY:
This trial is being conducted to evaluate the efficacy of Phasix™ Mesh implantation at the time of midline fascial closure compared to primary suture closure in preventing a subsequent incisional hernia in subjects at risk for incisional hernia after open midline laparotomy surgery.

DETAILED DESCRIPTION:
Subjects will be randomized (1:1) to one of the two treatment groups in the operating room after fascial closure.

ELIGIBILITY:
Inclusion Criteria:

1. Must be ≥ 18 years of age
2. Elective, open midline laparotomy ≥ 5 cm
3. Willing and able to provide written informed consent
4. Hernia risk equal to moderate or greater

Exclusion Criteria:

1. Previous hernia repair
2. Emergent surgery
3. Creation of skin flaps is preplanned
4. Preplanned 2nd surgery
5. Active skin pathology
6. Life expectancy less than 36 months
7. Pregnant or planning to become pregnant
8. Receiving a medication/medical condition that may adversely affect wound healing
9. ASA Class > IV
10. Enrolled in another clinical trial
11. Site personnel directly involved with this trial
12. Any condition that would preclude the use of the device or the subject form completing the follow-up requirements
13. Known or suspected allergy to tetracycline hydrochloride or kanamycin sulfate
14. Two separate incisions are created
15. Prior onlay mesh
16. Surgeon is unable to fully close the fascia
17. The surgery requires more than a single piece of mesh
18. Contraindication to placement of mesh
19. CDC Class IV/Active Infection
20. Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 477 (Estimated)
Dates: Start 2019-12-12 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Rate of Incisional Hernia | 36-Months
  The primary endpoint of the trial is the occurrence of incisional hernia in each treatment group (Phasix™ Mesh or Control Group)

SECONDARY OUTCOMES:
Rate of Incisional Hernia | 60-Months
  Rate of incisional hernia at each follow up time point
Rate of Device-related Adverse Events (AEs) | 60-Months
  Rate of Device-related Adverse Events (AEs)
Length of surgical procedure in minutes | Study Day 0
  Length of surgical procedure in minutes
Length of time for wound closure in minutes | Study Day 0
  Length of time for wound closure in minutes
Length of hospital stay in days | Through hospital stay, typically 3 days
  Length of hospital stay in days
Quality of Life: Optum Short Form Survey 12 Item Version 2 (SF-12v2®) | 60-Months
  Health-related quality of life will be measured using the Optum SF-12v2. The questionnaire consists of 12 items weighted and summed to provide physical and mental health scores from the subject's perspective (PCS and MCS). The two composite scores are computed using the scores on twelve questions that range from 0 to 100, with higher score indicating better quality of life.
Quality of Life: EuroQoL-5 Dimensions-3 Level (EQ-5D-3L©) | 60-months
  EuroQoL-Five Dimensions questionnaire-using Three Levels EQ-5D-3L is a standardized instrument for measuring generic health status. It consists of two components; health status description and evaluation. The health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression; each dimension ranging from 1-3. From these five dimensions, EQ-5D index is calculated, having a value between 0-1. The evaluation part involves visual analogue scale, asking the subject to mark health status on the day of the interview on a 20 cm vertical scale with end points of 0 and 100. Zero corresponds to " the worst health you can imagine", and hundred corresponds to "the best health you can imagine".

CONTACTS AND LOCATIONS:
Overall Officials: William Hope, MD, Principal Investigator — New Hanover Regional Medical Center
Locations (43):
- United States (30):
  - Dignity Health, Phoenix, Arizona
  - Keck Medical Center of USC, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - Hartford Hospital, Hartford, Connecticut
  - St. Francis Hospital and Medical Center, Hartford, Connecticut
  - Emory University, Atlanta, Georgia
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Kentucky Research Foundation, Lexington, Kentucky
  - Tulane University School of Medicine, New Orleans, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - Minneapolis VA Health Care System, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - St. Luke's Hospital, Kansas City, Missouri
  - Cox Health, Springfield, Missouri
  - Washington University, St Louis, Missouri
  - Nebraska Medical Center, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - New York Presbyterian Hospital-Columbia University Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Atrium Health, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - New Hanover Regional Medical Center, Wilmington, North Carolina
  - The Ohio State University, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Baptist Clinical Research Institute, Memphis, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - CAMC Health Education and Research Institute, Inc., Charleston, West Virginia
- Krankenhaus der Barmherzigen Brüder Graz, Graz, Austria
- Universitair Ziekenhuis Gent, Ghent, Belgium
- France (6):
  - CHU de Dijon Bourgogne, Dijon
  - Centre Hospitalier Universitaire de Lille, Lille
  - Hôpital Paris St Joseph, Paris
  - Hôpital Lyon Sud, Pierre-Bénite
  - CHU Reims, Reims
  - Hopitaux Universitaires de Strasbourg, Strasbourg
- Germany (5):
  - Charité - Universitätsmedizin Berlin, Campus Virchow Klinikum, Gyneocology, Berlin
  - Charité - Universitätsmedizin Berlin, Campus Virchow Klinikum, Surgery, Berlin
  - Asklepios Klinik Barmbek, Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Bundeswehrzentralkrankenhaus Koblenz, Koblenz

IPD SHARING:
Plan to Share IPD: No